CLINICAL TRIAL: NCT04435535
Title: Immediate Effects of Chest Physiotherapy in Tracheotomized Patients With Acute Respiratory Distress Syndrome.
Brief Title: Chest Physiotherapy in Tracheotomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jenny Örman, Physiotherapist, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEPpåtrack
Record Dates: First submitted 2020-06-02; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Breathing exercises; Intensive care; Physical therapy modalities; Physiotherapy; Respiratory distress syndrome, adult; Ventilator weaning
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive expiratory pressure (PEP) (Other): PEP 10 cmH2O 15 min
  Interventions: Procedure: PEP

INTERVENTIONS:
Procedure: PEP — Positive expiratory pressure 10 cmH2O 15 min

SUMMARY:
Positive expiratory pressure (PEP) breathing is common for treatment of different lung diseases and can increase lung volume and increase elimination of secretion from the airways. Today there is no evidence whether the treatment is effective or not for patients in the intensive care unit. The purpose of this study is to evaluate if PEP breathing can increase oxygenation for patients in the intensive care unit during weaning from the ventilator after acute respiratory distress syndrome.

PEP breathing will be applied on the tracheal cannula for 15 minutes. Measure of the PEP effect will be done before, during and for 20 minutes after PEP breathing.

DETAILED DESCRIPTION:
Procedure:

To achieve steady state, all subjects are positioned in a semi-recumbent position (30°) for 60 minutes before the start of the intervention and remain in that position during the entire investigation. Subjects are instructed to avoid talking and movements during both steady state and measurements. Airway suctioning (up to 20 kPa) through the tracheal cannula is performed only if there is risk for tube obstruction or if SpO2 decreases below 90%. Frequency of airway suctioning, and number of coughs during the study time are registered. An extra pre-intervention measurement is performed 15 minutes after the first to increase the validity of baseline measurements and control for changes in measured variables due to spontaneous variations.

A PEP device consisting of a one-way valve and exchangeable resistance nipples is used during the PEP breathing treatment. The resistance nipple is chosen at the start of the intervention aiming at an airway pressure of 10-15 cmH2O during tidal breathing (measured with a calibrated manometer). The duration of the PEP treatment is 15 minutes. Complementary oxygen is delivered at the same amount as before the intervention.

Measurements:

The primary outcome is PaO2. Five separate arterial blood samples of 0.7-1.5 ml each (altogether 3.5-7.5 ml for each subject) are drawn from an existing arterial catheter in the radial artery in the left or the right arm by nurses at the ward, and directly analysed.

Subject characteristics are registered from the clinical records, including gender, age, body mass index (BMI), smoking history, duration of invasive ventilation, and length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Tracheostomized participants
* ≥18 years old
* Moderate or severe ARDS during the ICU period, according to the Berlin definition.
* Ability to maintain PaO2 ≥ 67.5mmHg, with supplementary oxygen if needed, during spontaneous breathing for at least three consecutive hours.
* Normal curvature of the spine.

Exclusion Criteria:

* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change in PaO2 | Baseline. At 7 minutes and 15 minutes of intervention and 20 minutes post intervention.
  Change from baseline arterial partial pressure of oxygen

SECONDARY OUTCOMES:
Change in PaCO2 | Baseline. At 7 minutes and 15 minutes of intervention and 20 minutes post intervention.
  Change from baseline arterial partial pressure of carbon dioxide
Change in peripheral oxygen saturation (SpO2) | Baseline. At 7 minutes and 15 minutes of intervention and 20 minutes post intervention.
  Change from baseline in SpO2
Change in respiratory frequency | Baseline. At 7 minutes and 15 minutes of intervention and 20 minutes post intervention.
  Change from baseline in respiratory frequency
Change in mean arterial pressure (MAP) | Baseline. At 7 minutes and 15 minutes of intervention and 20 minutes post intervention.
  Change from baseline in MAP
Change in heart rate | Baseline. At 7 minutes and 15 minutes of intervention and 20 minutes post intervention.
  Change from baseline in heart rate
Change in Borg´s Category Ratio 10scale (Borg CR 10 scale) from baseline | Baseline. At 7 minutes and 15 minutes of intervention and 20 minutes post intervention.
  Borg CR-10 scale is an eleven point nominal scale that measures patient perceived breathlessness. A higher number indicates a greater breathlessness. 0=no breathlessness. 10 = very very high breathlessness (almost maximal).